CLINICAL TRIAL: NCT03933605
Title: Comparison of Palonosetron With Combined Palonosetron and Midazolam for Preventing Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Brief Title: Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Eun Kyung Choi, Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YUMC 2017-04-030
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Nausea; Postoperative Vomiting
Keywords: postoperative nausea and vomiting; midazolam; palonosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midazolam and palonosetron (Active Comparator): 0.05 mg/kg of midazolam i.v. with 0.075 mg of palonosetron i.v. was administered after anesthetic induction
  Interventions: Drug: midazolam and palonosetron group
- palonosetron (Active Comparator): the same volume (0.05 mg/kg) of normal saline i.v. with 0.075 mg of palonosetron i.v. was administered after anesthetic induction
  Interventions: Drug: palonosetron group

INTERVENTIONS:
Drug: midazolam and palonosetron group — intravenous midazolam and palonosetron administraion as prevention of postoperative nausea and vomiting
  Arms: midazolam and palonosetron
Drug: palonosetron group — intravenous palonosetron administraion as prevention of postoperative nausea and vomiting
  Arms: palonosetron

SUMMARY:
In the present study, midazolam and palonosetron in combination were more effective than palonosetron alone in lowering the incidence and severity of postoperative nausea and vomiting in the initial 2 h after laparoscopic cholecystectomy. Postoperative clinical complications were not different in both groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients (aged 20 to 65 years) scheduled for laparoscopic cholecystectomy with American Society of Anesthesiologists (ASA) physical status classification of 1 or 2

Exclusion Criteria:

* The patients with a history of allergy to any other drugs used in this study, gastrointestinal disorder, previous PONV, pregnant woman, breastfeeding woman, use of antiemetics within 24 hours or body mass index > 30 kg/m2

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | 24 hours after surgery
  0=none; 1=occur
severity of postoperative nausea and vomiting | 24 hours after surgery
  0 = absent; 1 = mild; 2 = moderate; 3 = severe

CONTACTS AND LOCATIONS:
Locations (1):
- Eun kyung Choi, Daegu, Korea (the Republic Of), South Korea

IPD SHARING:
Plan to Share IPD: Yes